CLINICAL TRIAL: NCT00823134
Title: Evaluation of ApneaLink Plus Scoring Capabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D2231-109
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-03

CONDITIONS: Sleep Apnea, Central; Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Central; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AL + polysomnography (Other): Participant wears an Apnea Link sleep apnoea screening device during the polysomnography to detect apnoeas (obstructive, central).
  Interventions: Device: ApneaLink Plus

INTERVENTIONS:
Device: ApneaLink Plus — Device used to evaluate for the presence of obstructive, central or mixed apneas
  Other Names: AL Plus

SUMMARY:
The purpose of this study is to investigate the following topics:

* Determine the accuracy of ApneaLink Plus in separating Apneas into Obstructive Apneas, Mixed Apneas and Central Apneas.
* Determine the accuracy of ApneaLink Plus in scoring Hypopneas according to the 2008 guidelines of the AASM = American Academy of Sleep Medcine.
* Determine whether patients can start and stop the recorder and are able to attach the additional effort sensor by themselves using the patient instruction sheet

DETAILED DESCRIPTION:
* Determine the accuracy of ApneaLink Plus in separating Apneas into Obstructive Apneas, Mixed Apneas and Central Apneas.
* Determine the accuracy of ApneaLink Plus in scoring Hypopneas according to the 2008 guidelines of the AASM = American Academy of Sleep Medcine.
* Determine whether patients can start and stop the recorder and are able to attach the additional effort sensor by themselves using the patient instruction sheet

ELIGIBILITY:
Inclusion Criteria:

* Willing to give written informed consent
* Adult patients who are 18 years of age or older
* No alcohol consumption 12 hrs before and during the trial period
* Normally sleep more than 3 hours per night

Exclusion Criteria:

* Unable to comprehend written and spoken German.
* Pregnant
* Patients who use of Bilevel PAP or CPAP therapy during the PSG
* Unsuitable for inclusion in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Knut Joechle, PhD, Study Director — ResMed; Heribert Knape, MD, Principal Investigator — Medizinische Klinik für Atemwegserkrankungen und Allergien, Fachkliniken Wangen
Locations (1):
- Medizinische Klinik für Atemwegserkrankungen und Allergien, Fachkliniken Wangen, Wangen, Baden-Wurttemberg, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- PSG/ApneaLink: Sleep Evaluation under Polysomnography and with ApneaLink
Period: Overall Study
Arm/Group | PSG/ApneaLink
Started | 23
Completed | 22
Not Completed | 1
Not completed — Invalid measurement | 1

BASELINE CHARACTERISTICS:
Arm/Group | PSG/ApneaLink
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.73 (16.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 22
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.77 (4.23)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Apnoea-Hypopnea-Index (Number of Apneas (All Apneas, Obstructive, Mixed, Central) and Number of Hypopneas) Between ApneaLink Plus and a PSG System Within the Same Evaluation Period
Description: Apnoea is defined as a decrease in flow of ≥90% from baseline for at least 10 seconds; hypopnea is a decrease in flow ≥30% from baseline for at least 10 seconds and an oxygen desaturation of ≥4%; obstructive: breathing efforts are ongoing; central: no breathing efforts
Time Frame: one night
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | PSG/ApneaLink
Number analyzed (Participants) | 22
events/hour
  AHI_psg | 14.77 (14.97)
  AHI_al | 12.14 (12.04)
Statistical Analysis 1: Comparison: PSG/ApneaLink; Test type: Other; p = 0.021, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2.8, Standard Deviation 4.7

2. Primary Outcome: Correlation Coefficient of Apnoea-Hypopnea-Index (AHI) (PSG) - AHI (AL)
Description: The AHI (PSG) values and AHI ApneaLink Plus (AL) value will be collected in one graph (Bland-Altmann Plot) and the correlation coefficient will be calculated. A correlation of >75% will be seen as threshold for validity.
Time Frame: 1 night
Population: Participant undergoes one night of sleep while wearing an Apnea Link device and polysomnography is being recorded.
Measure: Number; unit: correlation
Arm/Group | AL + Polysomnography
Number analyzed (Participants) | 22
correlation | 0.968
Statistical Analysis 1: Comparison: AL + Polysomnography; Per recording, the number of events found per category with PSG and ApneaLink Plus will be compared. As a summary, all PSG values and all ApneaLink Plus values per category will be collected in one graph (Bland-Altmann Plot). The correlation coefficient will be calculated per category. A correlation of >75% will be seen as threshold for validity; Test type: Other — The number of events found per category (PSG and ApneaLink Plus recording) will be compared. Events are Apneas and Hypopneas per hour of sleep, measured as Apnea-Hypopnea-Index (AHI), Apnea-Index (AI), Obstructive AI, Central AI, Hypopnea-Index (HI) and Oxygen Desaturation Index (ODI); Correlation coefficient (Bland-Altman) = 0.75

3. Primary Outcome: Correlation Coefficient of Apnoea-Index (AI) (PSG) - AI (AL)
Description: The AI (PSG) values and AI ApneaLink Plus (AL) value will be collected in one graph (Bland-Altmann Plot) and the correlation coefficient will be calculated. A correlation of >75% will be seen as threshold for validity.
Time Frame: 1 night
Population: Participant undergoes one night of sleep while wearing an Apnea Link device and polysomnography is being recorded.
Measure: Number; unit: Correlation
Arm/Group | AL + Polysomnography
Number analyzed (Participants) | 22
Correlation | 0.935

4. Primary Outcome: Correlation Coefficient of Obstructive-Apnoea-Index (OAI) (PSG) - OAI (AL)
Description: The OAI (PSG) values and OAI ApneaLink Plus (AL) value will be collected in one graph (Bland-Altmann Plot) and the correlation coefficient will be calculated. A correlation of >75% will be seen as threshold for validity.
Time Frame: 1 night
Population: Participant undergoes one night of sleep while wearing an Apnea Link device and polysomnography is being recorded.
Measure: Number; unit: Correlation
Arm/Group | AL + Polysomnography
Number analyzed (Participants) | 22
Correlation | 0.852

5. Primary Outcome: Correlation Coefficient of Central-Apnoea-Index (CAI) (PSG) - CAI (AL)
Description: The CAI (PSG) values and CAI ApneaLink Plus (AL) value will be collected in one graph (Bland-Altmann Plot) and the correlation coefficient will be calculated. A correlation of >75% will be seen as threshold for validity.
Time Frame: 1 night
Population: Participant undergoes one night of sleep while wearing an Apnea Link device and polysomnography is being recorded.
Measure: Number; unit: Correlation
Arm/Group | AL + Polysomnography
Number analyzed (Participants) | 22
Correlation | 0.939

6. Primary Outcome: Correlation Coefficient of Apnoea-Index (HI) (PSG) - HI (AL)
Description: The HI (PSG) values and HI ApneaLink Plus (AL) value will be collected in one graph (Bland-Altmann Plot) and the correlation coefficient will be calculated. A correlation of >75% will be seen as threshold for validity.
Time Frame: 1 night
Population: Participant undergoes one night of sleep while wearing an Apnea Link device and polysomnography is being recorded.
Measure: Number; unit: Correlation
Arm/Group | AL + Polysomnography
Number analyzed (Participants) | 22
Correlation | 0.754

7. Primary Outcome: Correlation Coefficient of Obstructive-Apnoea-Index (ODI) (PSG) - ODI (AL)
Description: The ODI (PSG) values and ODI ApneaLink Plus (AL) value will be collected in one graph (Bland-Altmann Plot) and the correlation coefficient will be calculated. A correlation of >75% will be seen as threshold for validity.
Time Frame: 1 night
Population: Participant undergoes one night of sleep while wearing an Apnea Link device and polysomnography is being recorded.
Measure: Number; unit: Correlation
Arm/Group | AL + Polysomnography
Number analyzed (Participants) | 22
Correlation | 0.905

ADVERSE EVENTS:
Arm/Group | PSG/ApneaLink
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No